CLINICAL TRIAL: NCT00750568
Title: Pharmacokinetics and Pharmacodynamics of Terbutaline Given as a Continuous Intravenous Infusion in Severe Status Asthmaticus
Brief Title: Intravenous Terbutaline in Severe Status Asthmaticus
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Wayne State University (Other)
Responsible Party: Kevin Valentine, MD, Children's Hospital of Michigan
Other Study IDs: 10904
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-08

CONDITIONS: Status Asthmaticus
Keywords: Bronchial asthma; Asthma, bronchial; Status Asthmaticus; Terbutaline sulfate
MeSH Terms: conditions — Status Asthmaticus; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: * In-patient in the Pediatric Intensive Care Unit
  * Diagnosis of Status asthmaticus
  * Receiving a continuous infusion of terbutaline as part of their standard of care
  * Ages 2 years to 6 years
- Group 2: * In-patient in the Pediatric Intensive Care Unit
  * Diagnosis of Status asthmaticus
  * Receiving a continuous infusion of terbutaline as part of their standard of care
  * Ages greater than 6 years to 12 years
- Group 3: * In-patient in the Pediatric Intensive Care Unit
  * Diagnosis of Status asthmaticus
  * Receiving a continuous infusion of terbutaline as part of their standard of care
  * Ages greater than 12 years to 18 years

SUMMARY:
Terbutaline is a medication that is used to treat serious asthma attacks (status asthmaticus). The purpose of this study is to determine if terbutaline is effective and safe when given as a continuous intravenous infusion to children ages 2 years to 18 years of age. Children participating in this study are inpatients in the Intensive Care Unit with a diagnosis of status asthmaticus and are receiving terbutaline as part of their routine care. Blood samples and physiological assessments will be used to determine how the body is using terbutaline and how well it is working.

DETAILED DESCRIPTION:
1. Background: Asthma remains a significant source of morbidity and mortality in children. In the United States, more than 11 million people reported having an asthma attack in the year 2000, and more than 5 percent of all children younger than age 18 reported having asthma attacks. The trend of increasing asthma-associated morbidity and mortality that occurred during 1980-1995 has not continued for all measures. During 1995-1998, the rate of emergency department visits for asthma increased, while the rate of hospitalization and death decreased for all age groups, except children younger than age 15. Asthma remains a significant problem despite scientific advances that generated greater understanding of the mechanisms of asthma and the development of therapeutic approaches that can reduce morbidity.

   Status asthmaticus is a common diagnosis for admission to pediatric intensive care units (PICUs). Widely accepted treatment for status asthmaticus includes inhaled beta-2 agonists, systemic corticosteroids, and inhaled anticholinergic agents. The intravenous and/or subcutaneous administration of beta-2 agonists has been advocated in the treatment of severe asthma and is prescribed in current practice. Additional treatment regimens may include magnesium, theophylline, and/or heliox with some patients still requiring mechanical ventilation, anesthetic agents or extracorporeal membrane oxygenation.

   Beta-adrenergic receptor agonists are critical in the treatment of asthma. Their use frequently results in effective bronchodilation. Commonly used beta-adrenergic agonists are epinephrine, albuterol and terbutaline, with albuterol and terbutaline having an increased selectivity for beta-2 receptors. These agents can be given by inhaled, IV, subcutaneous or oral routes. In the United States inhaled albuterol is the drug and route of choice in a majority of circumstances. Regarding efficacy when administering medications via the inhaled route, one must take into account many factors including inhalation technique, inspiratory flow rate, inspiratory volume and mode of delivery. Several characteristic pathophysiological changes that occur during a severe asthma attack (near complete airway obstruction, low tidal volumes, mucus plugging) may preclude the delivery of inhaled particles to the area of the lung that is most affected. In these instances, intravenous beta-agonists should be considered. Because of cardiac related side effects that are more pronounced in non-selective beta-agonist therapy, a beta-2 receptor agonist should be administered. In the United States, terbutaline is the only approved intravenous beta-2 receptor agonist.

   Terbutaline is a sympathomimetic amine synthesized in the mid-1960's that has been shown by in vitro and in vivo pharmacologic studies in animals to exert a preferential effect on beta 2-adrenergic receptors (beta2-AR), such as those located in bronchial smooth muscle. It has been available for clinical use since the 1970's and has been approved by the FDA for use in the treatment of asthma in children. Terbutaline binds to the beta-2 adrenergic receptor resulting in Gs-protein stimulation which in turn activates adenylyl cyclase increasing intracellular levels of 3'-5' cyclic adenosine monophosphate (cAMP). cAMP then activates protein kinase A (PKA) that phosphorylates several proteins that contribute to smooth muscle relaxation and resultant bronchodilation.
2. Hypothesis and Primary Objectives: Intravenous terbutaline by continuous infusion is effective in decreasing the severity of an acute asthma attack and is safe to use in children 2 years to 18 years old. Terbutaline has different pharmacokinetics when given by continuous infusion versus single dose administration.
3. Study Design: Phase 2 clinical pharmacokinetic/pharmacodynamic trial in pediatric patients aged 2-18 years old who are receiving intravenous terbutaline for a severe asthma attack. Three groups of 12 children will be examined based on age for a total N of 36. The first group will be 2-6 years, the second group will be 6-12 years old and the third will be adolescents 12-18 years old. Treatment efficacy will be gauged by comparing scores of the modified pulmonary index (MPIS) as well as utilization of the rescue medication protocol (see below). Pharmacokinetics and pharmacodynamics will be determined by serum samples collected in 1-2 ml aliquots prior to infusion and at 20 minutes, 2, 4, 6, 8, 10, and 12 hours post infusion, or until clinical improvement necessitates discontinuation of the infusion if less than 12 hours.
4. Study Components:

   * Modified Pulmonary Index Score (MPIS): Children will be assessed for clinical changes during therapy by utilizing the modified pulmonary index score (MPIS) which is a combination of 6 physiologic parameters, each graded 0-3, the sum of which reflects pulmonary status. The MPIS was assessed for reproducibility and validity and was shown to be highly reproducible across groups of health care providers (nurses, physicians, respiratory therapists) and was a valid indicator of asthma severity in children.
   * Terbutaline levels as determined by HPLC at designated times stated previously.

ELIGIBILITY:
Inclusion Criteria:

* Children 2 to 18 years of age.
* Admission to the ICU with a diagnosis of status asthmaticus.
* The pediatric intensivist taking care of the patient has decided to initiate intravenous terbutaline therapy.
* An indwelling venous catheter or arterial catheter that was placed for routine ICU monitoring.
* Informed consent obtained from the patient's parents or legal guardian.

Exclusion Criteria:

* Existing cardiovascular disease.
* History of bronchopulmonary dysplasia.
* Prior inclusion in this study.
* Known hypersensitivity to terbutaline, or prior adverse event associated with terbutaline.
* Terbutaline use within 48 hours of initiation of the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inpatients in Pediatric ICU with a diagnosis of status asthmaticus
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of continuous terbutaline infusion | Prior to infusion; 20 minutes, 2, 4, 6, 8, 10, 12 hours post infusion

SECONDARY OUTCOMES:
Modified Pulmonary Index Score (MPIS) | Assess every 4 hours while IV terbutaline is infusing, continuing for 8 hours after the infusion is discontinued
Physiologic parameters | Prior to terbutaline, 20 minutes post, then hourly during infusion
Side effects | Duration of continuous infusion

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Valentine, M.D., Principal Investigator — Children's Hospital of Michigan; Mary Lieh-Lai, M.D., Study Chair — Children's Hospital of Michigan; Wayne State University
Locations (3):
- United States (3):
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of Michigan, Detroit, Michigan
  - Rainbow Babies and Childrens' Hospital, Cleveland, Ohio